CLINICAL TRIAL: NCT01224210
Title: Ambrisentan in Patients With Porto-pulmonary Hypertension A Multicenter Open Label Trial
Acronym: Portopulm
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ambrisentan Portopulm Study
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Portopulmonary Hypertension
Keywords: portopulmonary hypertension; portal hypertension; esophageal or gastric varices; right heart catheterization; transpulmonary gradient; Endothelin Receptor Antagonist; Ambrisentan; Letairis; pulmonary hemodynamics
MeSH Terms: conditions — Hypertension, Portal; Esophageal and Gastric Varices | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ambrisentan (24 Weeks), Extension (4 Weeks) (Other): Open Label Ambrisentan
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — Ambrisentan once-daily in the morning with or without food. The adult dose selected for this study will be 5 mg for the first 4 weeks. After the initial 4 weeks the dose will be increased to 10mg (available doses are 5, and 10 mg) based on tolerance safety. Subjects will remain on 10mg until they complete the study. Dose adjustments may be made based on side effects.
  Other Names: Letairis

SUMMARY:
This is an Open Label, Multicenter, pilot clinical trial to assess the efficacy and safety of an oral selective Endothelin Receptor Antagonist (ambrisentan) in patients with portopulmonary hypertension.

Preliminary evidence suggests that ambrisentan is safe and effective in patients with portopulmonary hypertension. The goal of therapy for these patients is to improve symptoms of dyspnea and to improve pulmonary hemodynamics to a mean pulmonary artery pressure <35 mm Hg in order to make patients eligible for liver transplantation. Therefore, the primary endpoints for this study will include 6 minute walk distance (6MWD) and pulmonary vascular resistance (PVR).

Eligible subjects will receive 5 mg ambrisentan once-daily for the first 4 weeks. After the initial 4-week period, investigators will increase study drug dose to 10 mg once daily (both 5 mg and 10 mg doses are FDA approved). If 10 mg is not tolerated in the opinion of investigator, then the investigator may decrease the dose back to 5 mg once daily. Primary outcome is a change in both the 6 Minute Walk Distance and in Pulmonary Vascular Resistance from baseline to Week 24. Subjects will be monitored with liver function tests (LFT) every 2 weeks for the first 8 weeks, then every 4 weeks thereafter. These safety laboratory tests may be performed at a local phlebotomy laboratory or at the Investigator clinic. In addition, the Investigator will assess each subject for safety and efficacy at Week 4, Week 12, and Week 24. Following Week 24, subjects will be assessed for safety and efficacy every 12 weeks. Patients will be followed for a total of 1 year. After 1 year, if the Investigator feels that continuing the treatment will be beneficial to the patients, they will be provided with ambrisentan by Gilead Pharmaceuticals, free of charge.

ELIGIBILITY:
Inclusion Criteria:

Subjects need to fulfill all of the following 4 criteria:

1. Evidence of portal hypertension (by hemodynamic measurement, or by Doppler flow of portal circulation, or by clinical evidence of portal hypertension such as esophageal or gastric varices, as evidenced by prior upper endoscopy).
2. Evidence of pulmonary arterial hypertension by right heart catheterization (all three criteria need to be present) Right heart catheterization may have been performed up to 30 days prior to screening

   * Mean PAP (pulmonary artery pressure) >25 mm Hg, and
   * PVR (pulmonary vascular resistance) >240 dynes/s/cm5, and
   * TPG (transpulmonary gradient = meanPAP -PAWP) >12 mm Hg
3. Baseline AST, ALT < 5 times the upper limit of normal, total Bili < 3.0 mg/dl, and mild liver impairment with Child -Pugh class A or B
4. Ages 18 years and above

Exclusion Criteria:

1. Presence of any other etiology of pulmonary arterial hypertension (HIV, connective tissue disease, sickle cell, left heart failure, chronic thromboembolic PH, etc)
2. Treatment with prostacyclins, other ERAs, or PDE5 inhibitors within 30 days of enrollment.
3. Moribund state or anticipated death within 1 month.
4. AST or ALT ≥ 5 times upper limit of normal
5. Total bilirubin ≥ 3.0 mg/dl
6. Significant lung disease (obstructive lung disease with FEV1 < 1L, or FEV1/FVC <50%; or restrictive lung disease with Total Lung Capacity < 60% predicted). PFTs may have been performed up to 6 months prior to enrollment.
7. Pregnancy
8. Age <18 years
9. Child -Pugh class C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ioana Preston, MD, Principal Investigator — Tufts Medical Center
Locations (6):
- United States (6):
  - UCSD Medical Center, La Jolla, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Preston IR, Burger CD, Bartolome S, Safdar Z, Krowka M, Sood N, Ford HJ, Battarjee WF, Chakinala MM, Gomberg-Maitland M, Hill NS. Ambrisentan in portopulmonary hypertension: A multicenter, open-label trial. J Heart Lung Transplant. 2020 May;39(5):464-472. doi: 10.1016/j.healun.2019.12.008. Epub 2020 Jan 21. PMID 32008947

RESULTS

PARTICIPANT FLOW:
Groups:
- Ambrisentan (24 Weeks), Extension (4 Weeks): Treatment-naive Group 1 Pulmonary Arterial Hypertension patients with Porto-pulmonary Hypertension with Child-Pugh class A/B were administered with ambrisentan for 24 weeks, followed by a long-term extension (24-28 weeks).
Period: Overall Study
Arm/Group | Ambrisentan (24 Weeks), Extension (4 Weeks)
Started | 30
Completed | 23
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: Group 1 Pulmonary Arterial Hypertension with Porto-pulmonary Hypertension
Groups:
- Ambrisentan (24 Weeks), Extension (4 Weeks): Long-term extension of 24-28 weeks of ambrisentan.
Arm/Group | Ambrisentan (24 Weeks), Extension (4 Weeks)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19
pulmonary vascular resistance [Mean (Standard Deviation); unit: HRU/Wood units] | 7.1 (5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Vascular Resistance
Description: Change in Pulmonary Vascular Resistance from baseline to Week 24 for all patients (using cardiac output [CO] measured by the thermodilution method and reported as percent difference from baseline).
Time Frame: from baseline to Week 24
Measure: Mean (Standard Deviation); unit: percent difference from baseline
Groups:
- Ambrisentan: Open Label Ambrisentan
  Ambrisentan: Ambrisentan once-daily in the morning with or without food. The adult dose selected for this study will be 5 mg for the first 4 weeks. After the initial 4 weeks the dose will be increased to 10mg (available doses are 5, and 10 mg) based on tolerance safety. Subjects will remain on 10mg until they complete the study. Dose adjustments may be made based on side effects.
Arm/Group | Ambrisentan
Number analyzed (Participants) | 30
percent difference from baseline | 7.1 (5)

2. Primary Outcome: 6 Minute Walk Distance
Description: Change from baseline in 6 Minute Walk Distance to Week 24 for all patients. (difference measured in meters).
Time Frame: Change from baseline to Week 24
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Group 1 PAH With PoPH: Treatment-naive Group 1 PAH patients with PoPH with Child-Pugh class A/B were administered with ambrisentan for 24 weeks, followed by a long-term extension (24-28 weeks).
Arm/Group | Group 1 PAH With PoPH
Number analyzed (Participants) | 30
meters
  Baseline | 314 (94)
  Week 24 | 336 (108)

ADVERSE EVENTS:
Arm/Group | Ambrisentan (24 Weeks), Extension (4 Weeks)
All-Cause Mortality (participants affected / at risk) | 4/30
Serious Adverse Events (participants affected / at risk) | 14/30
Other Adverse Events (participants affected / at risk) | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambrisentan (24 Weeks), Extension (4 Weeks) (N=30)
Edema (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Headache (Musculoskeletal and connective tissue disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambrisentan (24 Weeks), Extension (4 Weeks) (N=30)
Leg Edema (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Standardization of the 6 Minute Walk Test

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No